CLINICAL TRIAL: NCT03359330
Title: A Multi-center Study on Mid-term Effect Observation of Biodegradable Conduit Small Gap Tublization Repairing Peripheral Nerve Injury
Brief Title: Mid-term Effect Observation of Biodegradable Conduit Small Gap Tublization Repairing Peripheral Nerve Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Peixun, Department of orthopaedics and trauma, Peking University People's Hospital
Other Study IDs: PKUPH-PNI
Record Dates: First submitted 2017-11-26; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Peripheral Nerve Injuries
Keywords: Peripheral nervous system diseases; Wounds and injuries; Nerve regeneration; Biocompatible materials; Surgical procedures
MeSH Terms: conditions — Peripheral Nerve Injuries; Peripheral Nervous System Diseases; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Degradable conduit small gap tublization: patients with fresh peripheral nerve injury in the upper extremities,repaired with degradable conduit small gap tublization
  Interventions: Other: Degradable Conduit Small Gap Tublization

INTERVENTIONS:
Other: Degradable Conduit Small Gap Tublization — Degradable Conduit Small Gap Tublization Repairing Peripheral Nerve Injury

SUMMARY:
To observe the Mid-term clinical effect of biodegradable conduit small gap tublization to repair peripheral nerve injury in multi-center．

DETAILED DESCRIPTION:
In the study，150 cases of fresh peripheral nerve injury in the upper extremities are recruited in multi-center． After formally informed and obtaining the consent，the biodegradable conduit small gap tublization are used to repair the nerve．Their nerve functional recovery conditions are clinically observed according to the standard score methods provided by SHEN Ning-jiang and British Medical Research Council at 3 years after surgery．The excellent and good rates of the overall nerve functional recovery are calculated．

ELIGIBILITY:
Inclusion Criteria:

* fresh peripheral nerve injury in the upper extremities

Exclusion Criteria:

* acute myocardial infarction history within 6 months,
* old and pathological peripheral nerve injury,
* acute and chronic infection,
* various consumptive diseases
* unable to tolerate surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with fresh peripheral nerve injury in the upper extremities, requiring surgery
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Nerve function 1 | 3 years after surgery
  standard score methods provided by British Medical Research Council

SECONDARY OUTCOMES:
Nerve function 2 | 3 years after surgery
  standard score methods provided by Shen Ningjiang Using MSA system

CONTACTS AND LOCATIONS:
Overall Officials: Peixun Zhang, MD, Principal Investigator — Department of orthopaedics and trauma

IPD SHARING:
Plan to Share IPD: No